CLINICAL TRIAL: NCT07198139
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of CDI-988 in Healthy Adults After Challenge With Norovirus
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics of CDI-988 in Healthy Adults After Challenge With Snow Mountain Virus
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDI-988-P1b-001
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Norovirus
Keywords: tolerability; viral challenge model; antiviral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Snow Mountain Virus (Other): Challenge with Snow Mountain Virus
  Interventions: Other: Snow Mountain Virus
- Stage 2: Drug CDI-988 (Experimental)
  Interventions: Drug: CDI-988; Other: Snow Mountain Virus
- Stage 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Snow Mountain Virus

INTERVENTIONS:
Drug: CDI-988 — Antiviral to treat norovirus
  Arms: Stage 2: Drug CDI-988
Drug: Placebo — Matching placebo
  Arms: Stage 2: Placebo
Other: Snow Mountain Virus — Challenge with Snow Mountain Virus

SUMMARY:
Participants in this study will be given either CDI-988 or placebo orally before receiving a norovirus challenge virus and continuing for 5 days. Participants will not know whether they are getting placebo or CDI-988. The study will evaluate how well CDI-988 compared to placebo can reduce the incidence of clinical symptoms after a challenge with norovirus. The amount of virus in stool samples will be measured over time. Side effects and pharmacokinetics (the amount of CDI-988 in blood) will also be measured.

DETAILED DESCRIPTION:
This is a single center Phase 1b randomized, double-blind, placebo-controlled study. The primary objective will be to evaluate the efficacy of CDI-988 in comparison to placebo in reducing the incidence of clinical symptoms after challenge with norovirus. Secondary objectives will be to evaluate the efficacy of CDI-988 in comparison to placebo in reducing viral shedding and disease severity and to evaluate the safety of CDI-988 in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female
* Aged 18 to 49 years
* Good state of health
* Known fucosyl transferase 2 (FUT2) secretor status

Exclusion Criteria:

* History of participation in any norovirus challenge or vaccine clinical trial
* Receipt or planned receipt of any non-live vaccines within 7 days or live vaccines within 30 days before screening or prior to Day 28
* History of suspected norovirus gastroenteritis or chronic/recurrent gastrointestinal symptoms (e.g., diarrhea or vomiting) within 2 years prior to screening
* History of diagnosed gastrointestinal malabsorption disorders, major gastrointestinal surgery, or diagnosed chronic GI conditions
* Presence of moderate or severe illness, fever (≥38°C), or diarrhea/vomiting within 7 days prior to challenge
* Any acute illness on Day 1 (dosing day)
* Positive Day 0 stool tests for enteric pathogens
* Body weight <45 kg or BMI <18 or >32 kg/m² on Day 0
* Use of immunosuppressive therapy within 6 months prior to Day 0 or having any primary or secondary immunocompromising condition
* Use of high-dose systemic corticosteroids (≥20 mg/day prednisolone for ≥2 weeks) or high-dose inhaled steroids for >7 days within 6 months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of norovirus-confirmed disease | Day 0 to Day 21
  Disease is defined as diarrhea and/or vomiting (during the inpatient period), with laboratory-confirmed infection (with SMV specific primers on stool/emesis) or seroconversion

SECONDARY OUTCOMES:
Modified Vesikari Score (MVS) symptom scores during the inpatient period in infected patients | Day 1 to Day 6
  Score based on duration of diarrhea, maximum number of stools in a 24 hour period, duration of vomiting and maximum number of vomiting episodes in a 24 hour period
Time to symptom improvement | Day 1 to Day 6
  From peak Total Symptom Score to point where Total Symptom Score is within 3 points of baseline prior to challenge. The Modified Vesikari Score is a clinical tool used to assess the severity of acute gastroenteritis in children. The minimum and maximum values are 0 and 20, respectively. Higher scores mean a worse clinical severity. For example, a higher score reflects more severe symptoms such as longer duration or higher frequency of diarrhea or vomiting.
Time to first SMV-negative stool | Day 1 to Day 6
  Determined by RT-qPCR
Area Under the Curve of SMV load | Day 1 to Day 21
  Determined by RT-qPCR
Incidence of treatment emergent adverse events | Day 0 to Day 21
  Number of participants with adverse events following first dose
Incidence of serious adverse events | From signing informed consent to Day 21
  Number of participants with serious adverse events
Maximum plasma concentration of CDI-988 | Day 0 and Day 4 pre-dose and at 2, 3, 4, 6, 8, and 12 hours
  Amount of CDI-988 in the blood
Time of maximum plasma concentration of CDI-988 | Day 0 and Day 4 pre-dose and at 2, 3, 4, 6, 8, and 12 hours
  time to reach maximum plasma concentration
Area under the plasma concentration time curve | Day 0 and Day 4 pre-dose and at 2, 3, 4, 6, 8, and 12 hours
  Measurement of area under the plasma concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Hope Clinic of the Emory Vaccine Center
Locations (1):
- Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate participant data will be available from this study